CLINICAL TRIAL: NCT03340792
Title: Evaluation of the Physiological and Psychological Effects of Ambulation Training Utilizing an Exoskeleton Robot on Subjects With Spinal Cord Injury
Brief Title: Effects of Ambulation Training Utilizing an Exoskeleton Robot on Subjects With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Nai-Hsin Meng, Director, Department of Physical Medicine and Rehabilitation, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DMR-107-085
Record Dates: First submitted 2017-11-07; First posted 2017-11-14 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Spinal Cord Injuries
Keywords: Exoskeleton Device; Rehabilitation; Body composition; Quality of Life
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Exoskeleton robot ambulation training (Experimental): Ambulation training utilizing an exoskeleton robot
  Interventions: Device: Ambulation training utilizing an exoskeleton robot

INTERVENTIONS:
Device: Ambulation training utilizing an exoskeleton robot — Participants undergo 40 hours of ambulation training utilizing an exosksleton robot within 3 months.

SUMMARY:
The present study aims to investigate the effects of ReWalk exoskeleton robot training on various physiological and psychological parameters among subjects with spinal cord injury, including body composition and bone mineral mass, balance ability, bowel and bladder symptoms, severity of pain, psychological well-being, and quality of life. Ten patients with paraplegia caused by spinal cord injury will be recruited from the out-patient clinic of Department of Physical Medicine and Rehabilitation at the China Medical University hospital. All participants will undergo dual X-ray absorptiometry to evaluate the baseline bone mineral density. Eligible participants will then take ReWalk training sessions comprises of 3 x 1-hour sessions per week for 40 sessions. A comprehensive battery of outcome measures, including body composition and bone mineral mass, balance ability, bowel and bladder symptoms, severity of pain, psychological well-being, and quality of life, will be utilized for comparison after 40 sessions of ReWalk ambulation training.

DETAILED DESCRIPTION:
The loss of upright mobility has a profound effect on the health and quality of life for individuals with a spinal cord injury (SCI). The ReWalk exoskeleton is an FDA-cleared, wearable, computer-controlled exoskeleton robot that enables subjects with SCI to stand and walk using crutches to keep balance. China Medical University Hospital is the second hospital in Taiwan to acquire this relatively new rehabilitation robot. ReWalk exoskeleton not only helps the patients with paraplegia regain their ability to walk, previous studies also suggest that restoration of upright mobility may help mitigate the physical and psychological decline routinely experienced by individuals with SCI.

The present study aims to investigate the effects of ReWalk exoskeleton robot training on various physiological and psychological parameters among subjects with spinal cord injury, including body composition and bone mineral mass, balance ability, bowel and bladder symptoms, severity of pain, psychological well-being, and quality of life. Ten patients with paraplegia caused by spinal cord injury will be recruited from the out-patient clinic of Department of Physical Medicine and Rehabilitation at the China Medical University hospital. All participants will undergo dual X-ray absorptiometry to evaluate the baseline bone mineral density. Eligible participants will then take ReWalk training sessions comprises of 3 x 1-hour sessions per week for 40 sessions. The first 20 or so hours of training sessions focus on basic ReWalk skills, and the following training sessions focus on advanced ReWalk skills. A comprehensive battery of outcome measures, including body composition and bone mineral mass, balance ability, bowel and bladder symptoms, severity of pain, psychological well-being, and quality of life, will be utilized to obtain an in-depth overview and comparison of the treatment efficacy after 40 sessions of ReWalk ambulation training. The measures include: muscle strength measurements, Berg Balance Scale, modified Functional Reach Test, 10-Meters Walking Test, Timed Up and Go test, the Short Form-36 and Spinal Cord Injury-Quality Of Life questionnaires for health-related quality of life measurement. Dual X-ray absorptiometry will be used to measure the bone mineral density of the lumbar spine, the proximal femoral region and the distal forearms. It will also be used to estimate fat mass and lean body mass of the participants. All the outcome assessments, except for the Timed Up and Go and the 10-Metersr Walking Test, will be performed prior to the first training session and again at the end of the ReWalk ambulation training sessions. Descriptive data will be provided for all demographic parameters and with a mix-design ANOVA analysis employed to compare pre- and post-training conditions for all repeated outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Between the age of 20-65 years old;
2. Have paraplegia resulting from thoracic or lumbar spinal cord injury.
3. At least 6 months after onset of the spinal cord injury
4. Well motivated and willing to participate 40 hours of ReWalk ambulation training sessions.

Exclusion Criteria:

1. Have spinal cord injury neurologic level above T4
2. Height greater than 190 cm or lower than160 cm
3. Weight greater than 100 kg
4. Have osteoporosis (T-score < -2.5)
5. Deep vein thrombosis
6. Severe orthostatic hypotension precluding standing and walking training
7. Pregnancy
8. Cognitive impairments that would impact on the safe participation in the study
9. Severe spasticity of lower limbs (Modified Ashworth Scale >3)
10. Contracture of the ankle, or a knee flexion contracture greater than 10 degrees
11. Musculoskeletal conditions that affected gait capacity
12. Co-existence of other neurological diseases

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-11-23 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
bone mineral density | Change from baseline at 1 week after completion of 40 hours of ambulation training
  bone mineral density of the lumbar spine, the proximal femoral region and the distal forearms, measured by dual X-ray absorptiometry

SECONDARY OUTCOMES:
SF-36 | change from baseline at 1 week after completion of 40 hours of ambulation training
  SF-36 contains 36 items comprising eight subscales: physical functioning (PF), role limitations due to physical problems (RP), bodily pain, general health perceptions (GH), vitality (VT), social functioning (SF), role limitations due to emotional problems (RE), and mental health (MH). All subscales are transformed into a 0-100 scale, with 100 indicating the best status.
Spinal Cord Injury-Quality of Life measurement system | change from baseline at 1 week after completion of 40 hours of ambulation training
  The SCI-QOL consists of 19 item banks, including the SCI-Functional Index banks, and 3 fixed-length scales measuring physical, emotional, and social aspects of health-related QOL (HRQOL). A description of the score range (and which values are considered to be a better or worse outcome) is not included because it greatly exceeds the 999-character limitation allowed in the box of "descrpition"
  Emotional Health Domain:
  Positive Affect & Well-Being, Depression, Anxiety, Stigma, Resilience, Grief/Loss, Self-Esteem and Psychological Trauma
  Physical-Medical Health Domain:
  Skin/Pressure Ulcers Scale, Bladder Complications Scale, Bladder Management Difficulties, Bowel Management Difficulties, Pain Interference and Pain Behavior Scale.
  Social Participation Domain:
  Ability to Participate in Social Roles and Activities, Satisfaction with Social Roles and Activities, Independence.
  SCI-Functional Index banks: Basic Mobility, Ambulation, Fine Motor, Self-Care and Wheelchair activities.
fat mass | change from baseline at 1 week after completion of ambulation training
  fat mass measured by dual X-ray absorptiometry
lean body mass | change from baseline at 1 week after completion of 40 hours of ambulation training
  lean body mass measured by dual X-ray absorptiometry
Berg Balance Scale | change from baseline at 1 week after completion of 40 hours of ambulation training
  measuring sitting balance ability; minimum score: 0, maximu score 56; higher values represent a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Hsin Meng, M.D., Principal Investigator — China Medical University, China Medical University Hospital
Locations (1):
- China Medical University Hospial, Taichung, Taiwan